CLINICAL TRIAL: NCT04862975
Title: Pharmacokinetics of Antiretroviral Drugs in Lactating Women and Breastmilk Fed Infants Under 6 Months of Age in Botswana
Acronym: BMS02
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00107262; HHSN275201800003I (Other Grant/Funding Number: NICHD)
Record Dates: First submitted 2021-04-23; First posted 2021-04-28 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Lactating Women on Select DOI; Breastmilk Fed Infants of Mothers on Select DOI; HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — dolutegravir; Lamivudine; Emtricitabine; Tenofovir

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Leftover specimens will be sent to the National Institutes of Child Health and Human Development (NICHD) repository for unknown future use.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Drug of Interest: Lactating moms receiving one or more antiretroviral drugs and their breastmilk fed infants per standard of care.
  Interventions: Drug: Dolutegravir; Drug: Lamivudine; Drug: Emtricitabine; Drug: Tenofovir Disoproxil Fumarate

INTERVENTIONS:
Drug: Dolutegravir — Dolutegravir will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider. Not prescribed for this study.
  Other Names: Dolutegravir Sodium; DTG
Drug: Lamivudine — Lamivudine will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider. Not prescribed for this study.
  Other Names: 3TC
Drug: Emtricitabine — Emtricitabine will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider. Not prescribed for this study.
  Other Names: FTC
Drug: Tenofovir Disoproxil Fumarate — Tenofovir Disoproxil Fumarate will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider. Not prescribed for this study.
  Other Names: Tenofovir DF; TDF

SUMMARY:
The purpose of this study is to characterize the pharmacokinetics (PK) of understudied drugs administered to lactating women, receiving antiretroviral drugs per SOC as prescribed by their healthcare provider, and their co-enrolled infants ≤180 days of age who receive maternal breastmilk.

DETAILED DESCRIPTION:
Prospective, single-site, open label, PK and safety study. Co-enrollment of lactating women ≥18 years of age receiving drugs of interest (DOIs) per standard of care (SOC), as prescribed by their healthcare providers, and their infants who receive maternal breastmilk ≤180 days postpartum.

To understand drug transfer into breastmilk and determine subsequent infant exposure, biological samples will be collected from lactating women (blood and breastmilk) and infants (blood). The opportunistic design of this study will allow for a minimal risk study, an expanded enrollment net, evaluation of antiretroviral drugs, and capitalization of procedures performed per SOC to maximize study efficiency and data collection and minimize potential risk to participants. The data collected through this initiative will provide valuable PK, dosing, and safety information for drugs in this vulnerable population in order to inform public health.

ELIGIBILITY:
Inclusion Criteria Mothers/Infants:

1. Lactating women ≥18 years of age who are receiving at least one DOI per SOC who are ≤180 days postpartum, and their infants (≤180 days of age) who receive maternal breastmilk.
2. Informed consent, according to local IRB/REB/IEC guidelines, prior to any study-related procedures.
3. If the mother is receiving more than one DOI, the mother must have taken all DOIs that she is receiving concomitantly for the 6 doses prior to sample collection.
4. Mother participant is fluent in English or Setswana.
5. Willing to provide at least 1 of the below required samples between the co-enrolled mother/infant pair:

   * Maternal breastmilk
   * Infant blood

Exclusion Criteria Mothers/Infants:

1. Any concomitant condition which, in the opinion of the participant's healthcare provider, the site principal investigator (PI), a research nurse, or designee conducting the study, would preclude participation in the study.
2. Known pregnancy of mother during sample collection.
3. Mother has pumped any breastmilk at all in between the last 6 direct infant feedings prior to sample collection.
4. Infant was fed breastmilk in any manner besides nursing at mother's breast for any of the last 6 feedings prior to sample collection.
5. Previous enrollment on this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 50 eligible lactating women and their breastmilk fed infants per DOI will be co-enrolled. Participants may be enrolled for one or more DOIs with a single consent. The co-enrollment of mothers and more than 1 infant (multiple birth) is permitted.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Drug concentration in maternal plasma | Baseline
  Drug concentration of a DOI in maternal plasma
Drug concentration in maternal breastmilk | Baseline
  Drug concentration of a DOI in maternal breastmilk
Drug concentration in infant plasma | Baseline
  Drug concentration of a DOI in infant plasma
Milk/Plasma ratio | Baseline
  The drug exposure of selected DOIs will be evaluated using milk/plasma ratio
Estimated daily infant dose | Baseline
  The drug exposure of selected DOIs will be evaluated using the estimated daily infant dose
Relative infant dose | Baseline
  The drug exposure of selected DOIs will be evaluated using relative infant dose
Infant/maternal exposure ratio | Baseline
  The drug exposure of selected DOIs will be evaluated using infant/maternal exposure ratio

OTHER OUTCOMES:
PK of selected DOIs in lactating women and breastmilk fed infants as measured by Clearance (CL) or apparent clearance (CL/F). | Baseline
  Clearance (CL) or apparent clearance (CL/F)
PK of selected DOIs in lactating women and breastmilk fed infants as measured by volume of distribution (V) or apparent volume of distribution (V/F) | Baseline
  Volume of distribution (V) or apparent volume of distribution (V/F)
PK of selected DOIs in lactating women and breastmilk fed infants as measured by elimination Half-life (t1/2). | Baseline
  Elimination Half-life (t1/2)
PK of selected DOIs in lactating women and breastmilk fed infants as measured by absorption rate constant (ka). | Baseline
  Absorption rate constant (ka)
PK of selected DOIs in lactating women and breastmilk fed infants as measured by area under the curve (AUC). | Baseline
  Area under the curve (AUC)
PK of selected DOIs in lactating women and breastmilk fed infants as measured by elimination rate constant (kel). | Baseline
  Elimination rate constant (kel)
PK of selected DOIs in lactating women and breastmilk fed infants as measured by maximum concentration (CMAX). | Baseline
  Maximum concentration (CMAX)
PK of selected DOIs in lactating women and breastmilk fed infants as measured by time to reach maximum concentration (TMAX). | Baseline
  Time to reach maximum concentration (TMAX)
Correlation of PK parameters (drug concentration in maternal breastmilk) with maternal BMI | Baseline
  Correlation of drug concentration of each DOI in maternal breastmilk with maternal BMI
Correlation of PK parameters (drug concentration in maternal plasma) with maternal BMI | Baseline
  Correlation of drug concentration of each DOI in maternal plasma with maternal BMI
Correlation of PK parameters (drug concentration in infant plasma) with maternal BMI | Baseline
  Correlation of drug concentration of each DOI in infant plasma with maternal BMI
Correlation of PK parameters (milk/plasma ratio) with maternal BMI | Baseline
  Correlation of milk/plasma ratio of each DOI with maternal BMI
Correlation of PK parameters (estimated daily infant dose) with maternal BMI | Baseline
  Correlation of estimated daily infant dose of each DOI with maternal BMI
Correlation of PK parameters (relative infant dose) with maternal BMI | Baseline
  Correlation of relative infant dose of each DOI with maternal BMI
Correlation of PK parameters (infant/maternal exposure ratio) with maternal BMI | Baseline
  Correlation of infant/maternal exposure ratio for each DOI with maternal BMI
Safety ESIs for infants | Baseline
  Will be collected from the medical record at the time of sample collection

CONTACTS AND LOCATIONS:
Overall Officials: Matt Kelly, MD, Principal Investigator — Duke University; Kevin Watt, MD, Principal Investigator — University of Utah; Stephen Balevic, MD, Principal Investigator — Duke University; Angelique Boutzoukas, MD, Principal Investigator — Duke University
Locations (4):
- South Africa (4):
  - Botswana-UPenn Partnership, Botswana, Gaborone
  - Lesirane Clinic, Botswana, Gaborone
  - Mogoditshane Clinic KDC, Botswana, Gaborone
  - Old Naledi Clinic, Botswana, Gaborone

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed, information about the study, including de-identified study data, will be submitted to the NIH data repository (https://dash.nichd.nih.gov and referred to below as "DASH"). With NIH approval, the data submitted to DASH may be used by other researchers for future research. The study data submitted to DASH will be de-identified, meaning it will not include any information that can identify the participant. The study team may also share the de-identified study data with other researchers. When the participant's de-identified study data are provided to other researchers for the purposes of future research, it will be done without obtaining additional permission from the participant.
Time Frame: Data will be uploaded to the repository within 2 years of study completion. Biological samples will be stored indefinitely. If a participant decides to withdraw from the study, they will be instructed per the ICF to contact the site investigator. Study data and samples that have been recorded / collected prior to withdrawal will continue to be used, but no new data or samples will be collected.
Access Criteria: In order to have access, researchers have to complete a Data access request. NICHD will review the request and either approve or deny it. IRB approval must be obtained by the researcher to access the data.
URL: http://dash.nichd.nih.gov/

REFERENCES:
- [Background] Ip S, Chung M, Raman G, Trikalinos TA, Lau J. A summary of the Agency for Healthcare Research and Quality's evidence report on breastfeeding in developed countries. Breastfeed Med. 2009 Oct;4 Suppl 1:S17-30. doi: 10.1089/bfm.2009.0050. PMID 19827919
- [Background] Carpenter RG, Gardner A, Jepson M, Taylor EM, Salvin A, Sunderland R, Emery JL, Pursall E, Roe J. Prevention of unexpected infant death. Evaluation of the first seven years of the Sheffield Intervention Programme. Lancet. 1983 Apr 2;1(8327):723-7. doi: 10.1016/s0140-6736(83)92023-8. PMID 6132080
- [Background] Cunningham AS, Jelliffe DB, Jelliffe EF. Breast-feeding and health in the 1980s: a global epidemiologic review. J Pediatr. 1991 May;118(5):659-66. doi: 10.1016/s0022-3476(05)80023-x. PMID 2019919
- [Background] Ruiz-Palacios GM, Calva JJ, Pickering LK, Lopez-Vidal Y, Volkow P, Pezzarossi H, West MS. Protection of breast-fed infants against Campylobacter diarrhea by antibodies in human milk. J Pediatr. 1990 May;116(5):707-13. doi: 10.1016/s0022-3476(05)82652-6. PMID 2329419
- [Background] Koletzko S, Sherman P, Corey M, Griffiths A, Smith C. Role of infant feeding practices in development of Crohn's disease in childhood. BMJ. 1989 Jun 17;298(6688):1617-8. doi: 10.1136/bmj.298.6688.1617. No abstract available. PMID 2503151
- [Background] Mayer EJ, Hamman RF, Gay EC, Lezotte DC, Savitz DA, Klingensmith GJ. Reduced risk of IDDM among breast-fed children. The Colorado IDDM Registry. Diabetes. 1988 Dec;37(12):1625-32. doi: 10.2337/diab.37.12.1625. PMID 3192037
- [Background] Kramer MS, Aboud F, Mironova E, Vanilovich I, Platt RW, Matush L, Igumnov S, Fombonne E, Bogdanovich N, Ducruet T, Collet JP, Chalmers B, Hodnett E, Davidovsky S, Skugarevsky O, Trofimovich O, Kozlova L, Shapiro S; Promotion of Breastfeeding Intervention Trial (PROBIT) Study Group. Breastfeeding and child cognitive development: new evidence from a large randomized trial. Arch Gen Psychiatry. 2008 May;65(5):578-84. doi: 10.1001/archpsyc.65.5.578. PMID 18458209
- [Background] Huo D, Adebamowo CA, Ogundiran TO, Akang EE, Campbell O, Adenipekun A, Cummings S, Fackenthal J, Ademuyiwa F, Ahsan H, Olopade OI. Parity and breastfeeding are protective against breast cancer in Nigerian women. Br J Cancer. 2008 Mar 11;98(5):992-6. doi: 10.1038/sj.bjc.6604275. Epub 2008 Feb 26. PMID 18301401
- [Background] Lord SJ, Bernstein L, Johnson KA, Malone KE, McDonald JA, Marchbanks PA, Simon MS, Strom BL, Press MF, Folger SG, Burkman RT, Deapen D, Spirtas R, Ursin G. Breast cancer risk and hormone receptor status in older women by parity, age of first birth, and breastfeeding: a case-control study. Cancer Epidemiol Biomarkers Prev. 2008 Jul;17(7):1723-30. doi: 10.1158/1055-9965.EPI-07-2824. PMID 18628424
- [Background] Danforth KN, Tworoger SS, Hecht JL, Rosner BA, Colditz GA, Hankinson SE. Breastfeeding and risk of ovarian cancer in two prospective cohorts. Cancer Causes Control. 2007 Jun;18(5):517-23. doi: 10.1007/s10552-007-0130-2. Epub 2007 Apr 21. PMID 17450440
- [Background] Chasela CS, Hudgens MG, Jamieson DJ, Kayira D, Hosseinipour MC, Kourtis AP, Martinson F, Tegha G, Knight RJ, Ahmed YI, Kamwendo DD, Hoffman IF, Ellington SR, Kacheche Z, Soko A, Wiener JB, Fiscus SA, Kazembe P, Mofolo IA, Chigwenembe M, Sichali DS, van der Horst CM; BAN Study Group. Maternal or infant antiretroviral drugs to reduce HIV-1 transmission. N Engl J Med. 2010 Jun 17;362(24):2271-81. doi: 10.1056/NEJMoa0911486. PMID 20554982
- [Background] Shapiro RL, Hughes MD, Ogwu A, Kitch D, Lockman S, Moffat C, Makhema J, Moyo S, Thior I, McIntosh K, van Widenfelt E, Leidner J, Powis K, Asmelash A, Tumbare E, Zwerski S, Sharma U, Handelsman E, Mburu K, Jayeoba O, Moko E, Souda S, Lubega E, Akhtar M, Wester C, Tuomola R, Snowden W, Martinez-Tristani M, Mazhani L, Essex M. Antiretroviral regimens in pregnancy and breast-feeding in Botswana. N Engl J Med. 2010 Jun 17;362(24):2282-94. doi: 10.1056/NEJMoa0907736. PMID 20554983
- [Background] Gardiner SJ, Kristensen JH, Begg EJ, Hackett LP, Wilson DA, Ilett KF, Kohan R, Rampono J. Transfer of olanzapine into breast milk, calculation of infant drug dose, and effect on breast-fed infants. Am J Psychiatry. 2003 Aug;160(8):1428-31. doi: 10.1176/appi.ajp.160.8.1428. PMID 12900304
- [Background] Atkinson HC, Begg EJ. Prediction of drug distribution into human milk from physicochemical characteristics. Clin Pharmacokinet. 1990 Feb;18(2):151-67. doi: 10.2165/00003088-199018020-00005. PMID 2318008
- [Background] Panchaud A, Garcia-Bournissen F, Csajka C, Kristensen JH, Taddio A, Ilett KF, Begg EJ, Ito S. Prediction of infant drug exposure through breastfeeding: population PK modeling and simulation of fluoxetine exposure. Clin Pharmacol Ther. 2011 Jun;89(6):830-6. doi: 10.1038/clpt.2011.23. Epub 2011 Apr 27. PMID 21525869
- [Background] Koshimichi H, Ito K, Hisaka A, Honma M, Suzuki H. Analysis and prediction of drug transfer into human milk taking into consideration secretion and reuptake clearances across the mammary epithelia. Drug Metab Dispos. 2011 Dec;39(12):2370-80. doi: 10.1124/dmd.111.040972. Epub 2011 Sep 22. PMID 21940904
- [Background] Fleishaker JC. Models and methods for predicting drug transfer into human milk. Adv Drug Deliv Rev. 2003 Apr 29;55(5):643-52. doi: 10.1016/s0169-409x(03)00032-2. PMID 12706547
- [Background] Ito S, Koren G. A novel index for expressing exposure of the infant to drugs in breast milk. Br J Clin Pharmacol. 1994 Aug;38(2):99-102. doi: 10.1111/j.1365-2125.1994.tb04331.x. PMID 7981020
- [Background] Atkinson H, Begg EJ. Concentrations of beta-blocking drugs in human milk. J Pediatr. 1990 Jan;116(1):156. doi: 10.1016/s0022-3476(05)81674-9. No abstract available. PMID 1967306
- [Background] Begg EJ, Duffull SB, Saunders DA, Buttimore RC, Ilett KF, Hackett LP, Yapp P, Wilson DA. Paroxetine in human milk. Br J Clin Pharmacol. 1999 Aug;48(2):142-7. doi: 10.1046/j.1365-2125.1999.00992.x. PMID 10417489
- [Background] Wojnar-Horton RE, Kristensen JH, Yapp P, Ilett KF, Dusci LJ, Hackett LP. Methadone distribution and excretion into breast milk of clients in a methadone maintenance programme. Br J Clin Pharmacol. 1997 Dec;44(6):543-7. doi: 10.1046/j.1365-2125.1997.t01-1-00624.x. PMID 9431829
- [Background] Ohman I, Vitols S, Luef G, Soderfeldt B, Tomson T. Topiramate kinetics during delivery, lactation, and in the neonate: preliminary observations. Epilepsia. 2002 Oct;43(10):1157-60. doi: 10.1046/j.1528-1157.2002.12502.x. PMID 12366729
- [Background] Kobbe R, Schalkwijk S, Dunay G, Eberhard JM, Schulze-Sturm U, Hollwitz B, Degen O, Teulen M, Colbers A, Burger D. Dolutegravir in breast milk and maternal and infant plasma during breastfeeding. AIDS. 2016 Nov 13;30(17):2731-2733. doi: 10.1097/QAD.0000000000001259. No abstract available. PMID 27782968
- [Background] Gini J, Penchala SD, Amara A, Challenger E, Egan D, Waitt C, Lamorde M, Orrell C, Myer L, Khoo S, Else LJ. Validation and clinical application of a novel LC-MS method for quantification of dolutegravir in breast milk. Bioanalysis. 2018 Dec;10(23):1933-1945. doi: 10.4155/bio-2018-0085. Epub 2018 Nov 19. PMID 30450920
- [Background] Waitt C, Orrell C, Walimbwa S, Singh Y, Kintu K, Simmons B, Kaboggoza J, Sihlangu M, Coombs JA, Malaba T, Byamugisha J, Amara A, Gini J, Else L, Heiburg C, Hodel EM, Reynolds H, Mehta U, Byakika-Kibwika P, Hill A, Myer L, Lamorde M, Khoo S. Safety and pharmacokinetics of dolutegravir in pregnant mothers with HIV infection and their neonates: A randomised trial (DolPHIN-1 study). PLoS Med. 2019 Sep 20;16(9):e1002895. doi: 10.1371/journal.pmed.1002895. eCollection 2019 Sep. PMID 31539371
- [Background] Dickinson L, Kintu K, Coombs J, et al. Population pk of dolutegravir in plasma, cord, and breastmilk: results from DolPHIN-1. Presented at: Conference on Retroviruses and Opportunistic Infections 2019. Seattle, Washington. . 2019. https://www.croiconference.org/abstract/population-pk-dolutegravir-plasma-cord-and-breastmilk-results-dolphin-1/
- [Background] Mugwanya KK, Hendrix CW, Mugo NR, Marzinke M, Katabira ET, Ngure K, Semiyaga NB, John-Stewart G, Muwonge TR, Muthuri G, Stergachis A, Celum CL, Baeten JM. Pre-exposure Prophylaxis Use by Breastfeeding HIV-Uninfected Women: A Prospective Short-Term Study of Antiretroviral Excretion in Breast Milk and Infant Absorption. PLoS Med. 2016 Sep 27;13(9):e1002132. doi: 10.1371/journal.pmed.1002132. eCollection 2016 Sep. PMID 27676257
- [Background] Benaboud S, Pruvost A, Coffie PA, Ekouevi DK, Urien S, Arrive E, Blanche S, Theodoro F, Avit D, Dabis F, Treluyer JM, Hirt D. Concentrations of tenofovir and emtricitabine in breast milk of HIV-1-infected women in Abidjan, Cote d'Ivoire, in the ANRS 12109 TEmAA Study, Step 2. Antimicrob Agents Chemother. 2011 Mar;55(3):1315-7. doi: 10.1128/AAC.00514-10. Epub 2010 Dec 20. PMID 21173182
- [Background] Bierhoff M, Smolders EJ, Tarning J, Burger DM, Spijker R, Rijken MJ, Angkurawaranon C, McGready R, White NJ, Nosten F, van Vugt M. Pharmacokinetics of oral tenofovir disoproxil fumarate in pregnancy and lactation: a systematic review. Antivir Ther. 2019;24(7):529-540. doi: 10.3851/IMP3341. PMID 31868655
- [Background] Gouraud A, Millaret A, Bernard N, et al. Tenofovir exposure through breast feeding: Serum concentrations in neonates and clinical follow-up. Fundam Clin Pharmacol 2012;26 (Suppl 1):9.
- [Background] ViiV Healthcare Company. TIVICAY PD- dolutegravir sodium tablet, for suspension TIVICAY- dolutegravir sodium tablet, film coated [package insert]. U.S. Dept. of Health and Human Services, Food and Drug Administration. June 12, 2020.
- [Background] GlaxoSmithCline. EPIVIR-lamivudine tablets for oral use [package insert]. U.S. Dept. of Health and Human Services, Food and Drug Administration. September, 2017.
- [Background] GlaxoSmithCline. EPIVIR- lamivudine oral solution [package insert]. U.S. Dept. of Health and Human Services, Food and Drug Administration. September, 2017.
- [Background] AvKARE. TENOFOVIR DISOPROXIL FUMARATE- tenofovir disoproxil fumarate tablet, film coated [package insert]. U.S. Dept. of Health and Human Services, Food and Drug Administration. April 21, 2020.
- [Background] Mirochnick M, Thomas T, Capparelli E, Zeh C, Holland D, Masaba R, Odhiambo P, Fowler MG, Weidle PJ, Thigpen MC. Antiretroviral concentrations in breast-feeding infants of mothers receiving highly active antiretroviral therapy. Antimicrob Agents Chemother. 2009 Mar;53(3):1170-6. doi: 10.1128/AAC.01117-08. Epub 2008 Dec 29. PMID 19114673
- [Background] Waitt CJ, Garner P, Bonnett LJ, Khoo SH, Else LJ. Is infant exposure to antiretroviral drugs during breastfeeding quantitatively important? A systematic review and meta-analysis of pharmacokinetic studies. J Antimicrob Chemother. 2015 Jul;70(7):1928-41. doi: 10.1093/jac/dkv080. Epub 2015 Apr 8. PMID 25858354
- [Background] Davis NL, Corbett A, Kaullen J, Nelson JAE, Chasela CS, Sichali D, Hudgens MG, Miller WC, Jamieson DJ, Kourtis AP. Antiretroviral Drug Concentrations in Breastmilk, Maternal HIV Viral Load, and HIV Transmission to the Infant: Results From the BAN Study. J Acquir Immune Defic Syndr. 2019 Apr 1;80(4):467-473. doi: 10.1097/QAI.0000000000001941. PMID 30570527
- [Background] Aebi-Popp K, Kahlert CR, Crisinel PA, Decosterd L, Saldanha SA, Hoesli I, Martinez De Tejada B, Duppenthaler A, Rauch A, Marzolini C; Swiss Mother and Child HIV Cohort Study (SHCS). Transfer of antiretroviral drugs into breastmilk: a prospective study from the Swiss Mother and Child HIV Cohort Study. J Antimicrob Chemother. 2022 Nov 28;77(12):3436-3442. doi: 10.1093/jac/dkac337. PMID 36177836
- [Background] Dickinson L, Walimbwa S, Singh Y, Kaboggoza J, Kintu K, Sihlangu M, Coombs JA, Malaba TR, Byamugisha J, Pertinez H, Amara A, Gini J, Else L, Heiberg C, Hodel EM, Reynolds H, Myer L, Waitt C, Khoo S, Lamorde M, Orrell C; DolPHIN-1 Study Group. Infant Exposure to Dolutegravir Through Placental and Breast Milk Transfer: A Population Pharmacokinetic Analysis of DolPHIN-1. Clin Infect Dis. 2021 Sep 7;73(5):e1200-e1207. doi: 10.1093/cid/ciaa1861. PMID 33346335
- [Background] Mulligan N, Best BM, Wang J, Capparelli EV, Stek A, Barr E, Buschur SL, Acosta EP, Smith E, Chakhtoura N, Burchett S, Mirochnick M; IMPAACT P1026s Protocol Team. Dolutegravir pharmacokinetics in pregnant and postpartum women living with HIV. AIDS. 2018 Mar 27;32(6):729-737. doi: 10.1097/QAD.0000000000001755. PMID 29369162
- [Background] Waitt C, Olagunju A, Nakalema S, Kyohaire I, Owen A, Lamorde M, Khoo S. Plasma and breast milk pharmacokinetics of emtricitabine, tenofovir and lamivudine using dried blood and breast milk spots in nursing African mother-infant pairs. J Antimicrob Chemother. 2018 Apr 1;73(4):1013-1019. doi: 10.1093/jac/dkx507. PMID 29309634
- [Background] Palombi L, Pirillo MF, Marchei E, Jere H, Sagno JB, Luhanga R, Floridia M, Andreotti M, Galluzzo CM, Pichini S, Mwenda R, Mancinelli S, Marazzi MC, Vella S, Liotta G, Giuliano M. Concentrations of tenofovir, lamivudine and efavirenz in mothers and children enrolled under the Option B-Plus approach in Malawi. J Antimicrob Chemother. 2016 Apr;71(4):1027-30. doi: 10.1093/jac/dkv435. Epub 2015 Dec 17. PMID 26679247
- [Background] Palombi L, Pirillo MF, Andreotti M, Liotta G, Erba F, Sagno JB, Maulidi M, Ceffa S, Jere H, Marchei E, Pichini S, Galluzzo CM, Marazzi MC, Vella S, Giuliano M. Antiretroviral prophylaxis for breastfeeding transmission in Malawi: drug concentrations, virological efficacy and safety. Antivir Ther. 2012;17(8):1511-9. doi: 10.3851/IMP2315. Epub 2012 Aug 21. PMID 22910456
- [Background] Shapiro RL, Holland DT, Capparelli E, Lockman S, Thior I, Wester C, Stevens L, Peter T, Essex M, Connor JD, Mirochnick M. Antiretroviral concentrations in breast-feeding infants of women in Botswana receiving antiretroviral treatment. J Infect Dis. 2005 Sep 1;192(5):720-7. doi: 10.1086/432483. Epub 2005 Jul 27. PMID 16088821
- [Background] Corbett AH, Kayira D, White NR, Davis NL, Kourtis AP, Chasela C, Martinson F, Phiri G, Musisi B, Kamwendo D, Hudgens MG, Hosseinipour MC, Nelson JA, Ellington SR, Jamieson DJ, van der Horst C, Kashuba A; BAN Study Team. Antiretroviral pharmacokinetics in mothers and breastfeeding infants from 6 to 24 weeks post-partum: results of the BAN Study. Antivir Ther. 2014;19(6):587-95. doi: 10.3851/IMP2739. Epub 2014 Jan 24. PMID 24464632
- [Background] Hu X, Wang L, Xu F. Guides concerning tenofovir exposure via breastfeeding: A comparison of drug dosages by developmental stage. Int J Infect Dis. 2019 Oct;87:8-12. doi: 10.1016/j.ijid.2019.07.023. Epub 2019 Jul 26. PMID 31357055
- See also: UNICEF Botswana Key Demographic Indicators — http://data.unicef.org/country/bwa/
- See also: FDA: Clinical Lactation Studies: Considerations for Study Design Guidance for Industry — https://www.fda.gov/media/124749/download